CLINICAL TRIAL: NCT00074308
Title: A Phase I/II Study Of Imatinib Mesylate And Bevacizumab In Patients With Advanced Melanoma And Other Advanced Cancers
Brief Title: Imatinib Mesylate and Bevacizumab in Treating Patients With Advanced Melanoma or Other Advanced Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02564; 03903; CDR0000343804 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Results first posted 2018-01-16 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-05

CONDITIONS: Recurrent Melanoma; Stage III Melanoma; Stage IV Melanoma; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Melanoma | interventions — Imatinib Mesylate; Bevacizumab

ARMS (1):
- Arm I (Experimental): Patients receive oral imatinib mesylate once or twice daily on days 1-28 and bevacizumab IV over 30-90 minutes on days 1 and 14. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: imatinib mesylate; Biological: bevacizumab; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: imatinib mesylate — Given orally
  Other Names: CGP 57148; Gleevec; Glivec
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of combining imatinib mesylate with bevacizumab in treating patients who have advanced melanoma or other metastatic or unresectable cancer. Imatinib mesylate may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Bevacizumab may stop the growth of tumor cells by stopping blood flow to the tumor. Combining imatinib mesylate with bevacizumab may kill more tumor cells

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the tolerability, maximum tolerated dose, and lowest biologically active dose of imatinib mesylate and bevacizumab in patients with advanced melanoma or other advanced cancers.

II. Determine the response rate, time to progression, and survival of patients treated with this regimen.

III. Correlate clinical activity with inhibition of platelet-derived growth factor receptor beta, vascular endothelial growth factor receptor, flt-1, and markers of angiogenesis in patients treated with this regimen.

IV. Correlate clinical activity with alterations in tumor perfusion as assessed by dynamic contrast-enhanced MRI and Doppler ultrasound in patients treated with this regimen.

V. Correlate toxicity, clinical activity, and correlative endpoints with the steady-stage plasma concentration of imatinib mesylate in patients treated with this regimen.

OUTLINE: This is a dose-escalation, open-label study.

PHASE I (closed to accrual as of 8/23/04): Patients receive oral imatinib mesylate once or twice daily on days 1-28 and bevacizumab IV over 30-90 minutes on days 1 and 14. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of imatinib mesylate and bevacizumab until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PHASE II: Patients receive imatinib mesylate and bevacizumab as in phase I at the MTD.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of 1 of the following:

  * Metastatic or unresectable malignancy for which standard curative or palliative measures do not exist or are no longer effective (phase I) (phase I study closed to accrual as of 8/23/04)
  * Melanoma (phase I and II)
* Measurable disease (phase II)
* No history or clinical evidence of CNS disease, including primary brain tumor or brain metastases
* Performance status - ECOG 0-1
* More than 3 months
* WBC at least 3,000/mm^3
* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No history of bleeding diathesis or coagulopathy
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 2.5 times ULN
* INR no greater than 1.5
* APTT normal
* Creatinine no greater than 2.0 times ULN
* Creatinine clearance at least 40 mL/min
* No proteinuria
* Urinary protein less than 500 mg/24 hours
* No history of stroke
* No uncontrolled hypertension within the past 6 months

  * Blood pressure less than 150/100 mm Hg on a stable antihypertensive regimen
* None of the following within the past 6 months:

  * Myocardial infarction
  * Unstable angina
  * New York Heart Association class II-IV congestive heart failure
  * Serious cardiac arrhythmia requiring medication
  * Grade II or greater peripheral vascular disease
  * Transient ischemic attack
  * Cerebrovascular accident
  * Other arterial thromboembolic event
  * Other clinically significant cardiovascular disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for at least 3 months after study participation
* No seizures not controlled with standard medical therapy
* No prior allergic reactions attributed to Chinese hamster ovary cell products, other recombinant human antibodies, or compounds of similar chemical or biological composition to imatinib mesylate
* No serious, nonhealing wound, ulcer, or bone fracture
* No ongoing or active infection requiring parenteral antibiotics
* No significant traumatic injury within the past 28 days
* No psychiatric illness or social situation that would preclude study compliance
* No other concurrent uncontrolled illness
* More than 4 weeks since prior immunotherapy
* More than 8 weeks since prior monoclonal antibody therapy
* No concurrent prophylactic granulocyte or platelet colony-stimulating factors
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No more than 1 prior cytotoxic chemotherapy regimen for advanced disease (phase II)
* More than 4 weeks since prior radiotherapy
* More than 28 days since prior major surgical procedure or open biopsy
* Recovered from prior therapy
* No concurrent chronic daily aspirin (greater than 325 mg/day) or nonsteroidal anti-inflammatory drugs known to inhibit platelet function
* No recent or concurrent full-dose anticoagulants (except as required to maintain patency of preexisting permanent indwelling IV catheters) or thrombolytic agent
* No concurrent grapefruit juice
* No concurrent cytochrome P450 enzyme-inducing antiepileptic drugs (e.g., phenytoin, carbamazepine, or phenobarbital)
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational or commercial agents or therapies directed at the malignancy
* No other concurrent investigational agents

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Flaherty, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 - Dose 1: Bevacizumab (5 mg/kg) Imatinib (400 mg/day)
- Phase 1 Dose 2; Phase 2: Bevacizumab (10 mg/kg) Imatinib (400 mg/day)
- Phase 1 Dose 3: Bevacizumab (10 mg/kg) Imatinib (600 mg/day)
- Phase 1 Dose 4: Bevacizumab (10 mg/kg) Imatinib (800 mg/day)
Period: Overall Study
Arm/Group | Phase 1 - Dose 1 | Phase 1 Dose 2 | Phase 1 Dose 3 | Phase 1 Dose 4 | Phase 2
Started | 3 | 3 | 3 | 8 | 23
Completed | 3 | 3 | 3 | 8 | 23
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total of 40 patients were enrolled (Phase 1= 17; Phase 2 = 23)
Groups:
- Phase 1: Patients receive oral imatinib mesylate once or twice daily (400-800 mg/day) on days 1-28 and bevacizumab IV (5-10mg/kg) over 30-90 minutes on days 1 and 14. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase 2: Patients receive oral imatinib mesylate once or twice daily (400 mg/day) on days 1-28 and bevacizumab IV (10mg/kg) over 30-90 minutes on days 1 and 14. Courses repeat every 28 days in the absence of disease progression or unacceptance toxicity.
- Total: Total of all reporting groups
Arm/Group | Phase 1 | Phase 2 | Total
Number analyzed (Participants) | 17 | 23 | 40
Age, Categorical [Count of Participants; unit: Participants]
  Arm 1: <=18 years | 0 | 0 | 0
  Arm 1: Between 18 and 65 years | 17 | 23 | 40
  Arm 1: >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Arm 1: Female | 4 | 7 | 11
  Arm 1: Male | 13 | 16 | 29
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 23 | 40

OUTCOME MEASURES:

1. Primary Outcome: MTD, Defined as One Dose Level Below the Dose That Induced DLT in at Least One Third of Patients at a Dose Level, Graded According to NCI CTCAE Version 3.0 (Phase I)
Time Frame: Up to 28 days
Measure: Number; unit: dose level
Groups:
- Phase 1 = Dose Escalation: Patients receive oral imatinib mesylate once or twice daily on days 1-28 and bevacizumab IV over 30-90 minutes on days 1 and 14. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  imatinib mesylate: Given orally
  bevacizumab: Given IV
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
Arm/Group | Phase 1 = Dose Escalation
Number analyzed (Participants) | 17
dose level | 2

2. Primary Outcome: Progression-free Survival at 16 Weeks (Phase II)
Description: Progression Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2 = Dose Expansion: Patients receive oral imatinib mesylate once or twice daily on days 1-28 and bevacizumab IV over 30-90 minutes on days 1 and 14. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  imatinib mesylate: Given orally
  bevacizumab: Given IV
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
Arm/Group | Phase 2 = Dose Expansion
Number analyzed (Participants) | 23
Participants | 8

3. Secondary Outcome: Response Rate at 8 Weeks, Evaluated Using RECIST (Phase II)
Description: Response and progression was evaluated in this study using Response Evaluation Criteria in Solid Tumors (RECIST).
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 = Dose Expansion
Number analyzed (Participants) | 23
Participants | 1

4. Secondary Outcome: Overall Survival (Phase II)
Description: Kaplan-Meier estimates of overall survival and 95% confidence intervals will be calculated.
Time Frame: Up to 6 years
Population: Data not collected
Arm/Group | Arm I
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Grades 1 and 2 events are included as non-serious. Grade 3 and 4 events are included as serious
Arm/Group | Phase 1 - Dose 1 | Phase 1 Dose 2 | Phase 1 Dose 3 | Phase 1 Dose 4 | Phase 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/8 | 2/23
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 1/8 | 1/23
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 1/8 | 1/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 - Dose 1 (N=3) | Phase 1 Dose 2 (N=3) | Phase 1 Dose 3 (N=3) | Phase 1 Dose 4 (N=8) | Phase 2 (N=23)
Blood and lympathic system disorders (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Anemia
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea/vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal insufficiency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 - Dose 1 (N=3) | Phase 1 Dose 2 (N=3) | Phase 1 Dose 3 (N=3) | Phase 1 Dose 4 (N=8) | Phase 2 (N=23)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flushing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea/vomiting (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Weight gain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Weight loss (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anorexia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal insufficiency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less